CLINICAL TRIAL: NCT06207097
Title: Effect of Dry Needling Plus Exercise Compared to Elastic Taping Plus Exercise on the Reduction of Nonspecific Low Back Pain and Functionality
Brief Title: Compare the Effect of Exercise Program Plus Dry Needling Versus Elastic Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Ignacio Astudillo Ganora, PhD, University of Americas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEC_FP_2023022
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling plus exercise program. (Experimental)
  Interventions: Other: physiotherapy techniques
- Elastic taping plus exercise program. (Experimental)
  Interventions: Other: physiotherapy techniques

INTERVENTIONS:
Other: physiotherapy techniques — Dry neeling: invasive physiotherapy technique where an acupuncture needle is used on painful points Elastic taping: physiotherapy technique where elastic bandage is used on the skin Exercise program: physical exercise prescription

SUMMARY:
Low back pain is a common musculoskeletal health condition in society. It is a leading cause of disability globally and has created a significant burden in terms of work disability and high healthcare costs.

Studies on the treatment of combined therapies for non-specific low back pain are scarce, so it is not known in depth which intervention is the best for reducing pain. For this reason, the objective of this study was to evaluate and compare the effect of physical exercise plus dry needling versus physical exercise plus elastic bandage. For this, a randomized clinical trial was carried out with a total of 22 people, where pain was evaluated using the ENA scale and functionality using the Oswestry test. Participants received CORE stabilization exercises. CORE stability training has become a popular training trend and has begun to be applied in rehabilitation programs and sports medicine (1).

The expected results of the study are that the group that receives the physical exercise intervention plus dry needling will have better results in reducing the pain and functionality variable, evaluated with ENA and Oswestry in 4 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Workers of the University of the Americas, Santiago Centro Campus, Echaurren and República Headquarters

Exclusion Criteria:

Not having a diagnosis of cancer,

* Hernia of the nucleus pulposus with neural symptoms,
* Pregnant
* History of recent surgery (<6 months)
* History of tumor
* History of spinal fracture
* People with belonephobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Pain (pain scale (VAS) 1 to 109 | 1 week
  visual analog pain scale

SECONDARY OUTCOMES:
dysfunction (percentage of disability due to low back pain (from 0 to 10%)) | 1 week
  Evaluation of dysfunction due to low back pain with the Oswestry Dysfunction Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Astudillo, PhD, Principal Investigator — Universidad de las Americas
Locations (1):
- Universidad de las Americas, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No